CLINICAL TRIAL: NCT04553432
Title: Dry Eye OmniLenz Application of Omnigen Research Study
Acronym: DOORS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: NuVision (Unknown)
Responsible Party: Principal Investigator, James Wolffsohn, Professor of Optometry, Aston University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aston1612
Record Dates: First submitted 2020-09-04; First posted 2020-09-17 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Dry Eye
Keywords: dry eye disease; amniotic membrane; bandage contact lenses; symptoms; tear film stability; ocular surface damage
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: 1 month baseline followed by randomisation into treatment or control and 6 months follow-up
Who Masked: Participant, Investigator
Masking Description: Patient will not be aware whether bandage contact lens has an amniotic membrane beneath in periphery or not Masked investigator will perform the clinical examinations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omnigen + OmniLenz (Experimental): Omnigen amniotic membrane 17mm disk with 6mm central aperture place under 18mm OmniLenz bandage contact lens
  Interventions: Device: Amniotic membrane Omnigen[TM]; Device: Bandage soft Contact Lens OmniLenz[R]
- OmniLenz (Active Comparator): Bandage contact lens alone
  Interventions: Device: Bandage soft Contact Lens OmniLenz[R]

INTERVENTIONS:
Device: Amniotic membrane Omnigen[TM] — 17mm circular disk of processed amniotic tissue donated by mother after birth with a 6mm laser cut aperture to allow unimpeded vision https://www.nu-vision.co.uk/omnigen
  Arms: Omnigen + OmniLenz
Device: Bandage soft Contact Lens OmniLenz[R] — 18mm soft silicone-hydrogel contact lens https://www.nu-vision.co.uk/omnilenz

SUMMARY:
Dry eye disease (DED) is a disease of the ocular surface characterised by ocular surface inflammation and damage and neurosensory abnormalities. Tear film breakup leading to localised hyperosmolarity can result in ocular surface damage either directly or through the cascade of inflammation that it initiates. Transplantation of human amniotic membrane has been used for many ophthalmic indications including many related to inflammation of the ocular surface.

A recent study published by McDonald and colleagues in 2018 conducted in 84 DED patients (97 eyes) receiving cryopreserved AM treatment (Prokera) in addition to prior maximal medical management demonstrated an improved ocular surface along with a notable reduction in disease severity scores.

Omnigen is a dehydrated amniotic membrane derived from human sources and certified by the UK Human Tissue Authority. OmniLenz Bandage Contact Lens (BCL) is a bespoke bandage contact lens (BCL) designed to enable the application of Omnigen without the need for either sutures or glue. The application procedure takes approximately 15 minutes and the patients wear the lens continually. The McDonald study indicates that any improvement seen persists for at least three months.

This study aims to expand on the work by McDonald et al. The study will be a randomised, parallel group study comparing Omnigen treatment applied with an OmniLenz BCL to OmniLenz BCL alone. The later treatment enables a degree of masking and for any difference to be attributable to the Omnigen rather than a contact lens. This is in line with the recommendations laid out be the DEWS group. Interim data and analysis will be conducted after enrolment of 20 patients. Following the first week application the eye will be assessed, and a further treatment applied for a further week. Therefore, the total treatment period will be two weeks with follow-up assessments at one and three months. At six months patients will complete an OSDI and EQ-5D assessment via email or post. The primary efficacy variability will be change in OSDI score, a patient reported scoring of dry eye symptoms. A number of clinical assessments of the ocular surface will also be performed as part of the secondary outcomes whilst the opportunity to measure a number of exploratory measures will enable further work following this study.

DETAILED DESCRIPTION:
The TFOS DEWS II report redefines dry eye as:

". . . a multifactorial disease of the ocular surface characterised by a loss of homeostasis of the tear film, and accompanied by ocular symptoms, in which tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neurosensory abnormalities play etiological roles." Dry eye disease (DED) is a global problem, afflicting at least 344 million people worldwide, and is one of the most frequent causes of patient visits to eye care practitioners. However, the epidemiology of DED continues to be a challenge due to the lack of a standardised worldwide definition. The prevalence of DED, with and without symptoms, ranges from 5 to 50%.

Tear hyperosmolarity, as well as inflammatory mediators, may induce DED symptoms and cause damage to epithelial cells, surface microvilli, barrier function, the glycocalyx, and goblet cells. Epithelial cell damage, lipid layer and blinking abnormalities, defective glycocalyx, loss of gel mucin and reduction in tear volume may result in loss of lubrication between the globe and eyelids, resulting in increased friction and also symptoms.

Inflammation of the ocular surface can cause inhibition of lacrimal secretion and loss of epithelial barrier function at the ocular surface. Tear film breakup, leading to localised hyperosmolarity, can result in ocular surface damage either directly or through the cascade of inflammation that it initiates. Improved understanding of the role of subclinical inflammation in the early stages of DED also warrants further study.

Amniotic membrane (AM) has been utilised for many years as an adjuvant for tissue healing, with the first recorded use by Davis in 1910 during skin transplantation and in the 1930s by Sorsby for chemical injuries to the eye. Transplantation of human amniotic membrane has since been used for many ophthalmic indications. Reports describe its efficacy in reconstructing a corneal surface severely damaged by chemical agents, promoting the healing of persistent corneal epithelial defects, enhancing the success of corneal surface reconstruction surgery and substituting for conjunctival autografts after excision of pterygium or removal of conjunctival lesions.

Human AM has anti-bacterial, anti-angiogenic, anti-inflammatory and anti-fibroblastic properties. These characteristics may play a role in the use of AM in the treatment of DED. A recent study published by McDonald and colleagues in 2018 conducted in 84 patients (97 eyes) receiving cryopreserved AM treatment (Prokera) in addition to prior maximal medical management demonstrated an improved ocular surface along with a notable reduction of the severity of the overall DEWS score up to three months post treatment. Note the DEWS score is not a common assessment approach (as opposed to the OSDI score) but is indicative that amniotic membrane may have a positive effect in dry eye.

Omnigen is a dehydrated amniotic membrane derived from human sources and certified by the UK Human Tissue Authority. It offers significant potential benefits compared to cryopreserved AM such as the ability to store at room temperature and to create optimum application options such as circular discs rather than squares. More importantly, Omnigen has been demonstrated to preserve more of the biochemistry of AM during processing which in turn should yield improved clinical outcomes. Omnigen is licenced for human application and is regulated by the Human Tissue Authority (HTA). NuVision has delivered over 5,000 Omnigen treatments for Ophthalmology use, without any reports of adverse events (reporting a prerequisite of the HTA).

NuVision Biotherapies holds establishment licences under the HTA (Human Tissue Authority) that monitor and ensure the services and facilities comply with Good Manufacturing Practice. Many of the standard applied are above and beyond the minimum required by European/UK legislation and regulation. The donated tissue is collected aseptically in NHS operating theatres according to protocols approved by the HTA. These protocols include donor consent and testing, quarantine and release of product for clinical use. Once collected the donated tissue is processed in dedicated Grade A facilities and decontaminated using an antibiotic cocktail. The individual Omnigen pieces are also cut and packaged in controlled environments which are regularly assessed by the HTA. The final products are assessed through quality control procedures including individual visual examination and released only to units signing and applying the HTA approved tissue supply agreement. This enables full traceability from donor to patients.

During production individual Omnigen pieces are marked using a surgical pen with a logo that enables clinicians to determine correct orientation of Omnigen. For use with OmniLenz BCL the epithelial side of the tissue should be towards the ocular surface.

Omnigen pieces are individually packed in flat, sterile packaging. Each pack is clearly labelled according to HTA standards including individual item numbers in addition to batch details. The product is not irradiated and will remain sterile until opened. Omnigen is stored at room temperature which simplifies logistics. NuVision offer both advice and equipment to units receiving Omnigen but many units including the trial centre hold their own licences. This means they are also controlled and subject to inspection by the HTA. Enclosed within the packaging are adverse event or reaction reporting forms and advice that should such an event occur to telephone NuVision immediately. To date there are here are no reported cases of patient harm caused by the application of Omnigen.

OmniLenz is a bespoke BCL designed to enable the application of Omnigen without the need for either sutures or glue. OmniLenz BCL is a CE marked lens, modified from a standard lens produced by Menicon, that has been used to treat millions of people world-wide. The modifications are minor adjustment to the back geometry of the lens to allow OmniLenz BCL to be inserted over the amnion. This development has created the clinical opportunity to treat numerous clinical conditions with AM in an in-clinic environment, rather than a surgical setting. It has been designed to meet the needs of patients including comfort, aesthetics and transparency.

Over 900 in-clinic, suture less, applications of Omnigen using OmniLenz BCL have been used to date, predominantly for treatment of severe persistent epithelial defects and ocular inflammation conditions including DED.

The proposed DOORS study aims to examine the impact of applying Omnigen in the clinic without sutures, for patients suffering from moderate to severe DED. It aims in particular to examine the impact on both symptoms and pathology including Quality of Life (QoL) measurements and relevant clinical markers of disease progression. Of particular note is a measurement of tear film osmolarity, data of which is currently lacking in most studies to date.

The Ocular Surface Disease Index (OSDI), developed by the Outcomes Research Group at Allergan Inc (Irvine, Calif), is a 12-item questionnaire designed to provide a rapid assessment of the symptoms of ocular irritation consistent with dry eye disease and their impact on vision-related functioning.

Risks of treatment

Amniotic membrane is a human tissue and as such carries a risk of infection associated with receiving human tissue. These have been reduced at least by:

* Careful donor selection via medical assessment by trained clinical staff
* Infectious disease testing
* Omnigen is from donors who test negative for, Human immunodeficiency virus, Hepatitis B virus, Hepatitis C virus, Human T-lymphotropic virus 1 (HTLV-I), Syphilis, Cytomegalovirus
* Aseptic retrieval from living donors
* Processing in Grade A clean rooms
* Pathogen reduction by decontamination using an antibiotic cocktail during processing
* Quality control steps from donation through to final packaging performed by trained staff In particular, the risks of the use of any human tissue, or tissue derived product, must always consider the risk of prion infection. Prions are known to cause variant Creutzfeldt-Jakob disease (vCJD). CJD is a rare and fatal human degenerative condition which can be sporadic, inherited (familial), iatrogenic or variant. An analysis of all 177 UK vCJD cases reported up to December 2013 looking for the possibility of vCJD transmission through organ/tissue transplantation in the UK provided no evidence of transplant-associated vCJD in the UK. Therefore, this evidence suggests that previous UK factors as risk for CJD contamination are minimum to non-existent.

Omnigen is processed using the following antibiotics:

* Gentamycin 200 mg/ml
* Imipenem 10 mg/ml
* Nystatin 125,000 U/ml
* Polymyxin B 10 mg/ml
* Vancomycin 2.5 µg/ml Patients with antibiotic sensitivity should be identified and assessed according. Antibiotic levels in Omnigen are relatively low. When released from the tissue, most will be washed from the surface of the eye by tear production and blinking. However, research has shown that when drugs in tears come in contact with the vascular nasal mucosa, absorption into the bloodstream can occur. The 'one off' amount of antibiotic becoming systemic is unlikely to elicit and sensitivity reaction, but the potential risk needs to be considered.

Human amniotic membrane lacks immunogenicity, and the cornea has immune privilege. It is safe to say that over 1 million amniotic membrane transplantation procedures have been performed worldwide. However, there is no reported literature evidence of amniotic membrane eliciting an immune response at the ocular surface, even after repeat application from different donors. Therefore, though the potential risk still needs to be considered and explained to the patients, the risk of sensitivity is low. Where the patient is treated in the clinic using Omnigen, applied with OmniLenz BCL, the transplant can be rapidly removed should any response present itself.

Omnigen is processed using Raffinose a common lyoprotectant used in the preservation of cells and tissues, providing hypertonicity for cell desiccation. There is no reported literature evidence of any cases of sensitivity to raffinose pentahydrate.

The trial design has been selected to reflect the recommendations of Design and Conduct of Clinical Trials: Report of the Clinical Trials Subcommittee of the International Dry Eye WorkShop (2007). This stated that "the most desirable design of a clinical trial is a prospective, randomized, double-masked, placebo- or vehicle- controlled parallel group or crossover study".

The control arm has been chosen for the following reasons:

i) The intervention being studied comprises two elements; the intended amniotic membrane (Omnigen), and a modified bandage contact lens (OmniLenz BCL) which is used to hold the amnion in place but may have an indirect benefit. Therefore, any change may potentially be due to either element or a combination of both.

ii) The use of bandage contact lenses is a recognised treatment approach for DED. and represents an existing standard of care. OmniLenz BCL treatment alone is considered to be equivalent to a bandage contact lens.

iii) OmniLenz BCL placement will be obvious to the patient. The application of an OmniLenz BCL without Omnigen will enable the patient to remain masked to receiving the investigational intervention.

ELIGIBILITY:
Inclusion Criteria:

* A mean average score of 25 to 80 using more than one OSDI assessment in the last six weeks
* DED present for at least 12 months
* Informed consent
* Aged 18 or over on date of Baseline assessment
* Able to Attend Aston University
* No changes to current DED therapy in the last six weeks
* Presence of at least 1 of the following signs in the same eye at baseline visits

  * Corneal (≥5 punctate spots)
  * Conjunctival (≥9 punctate spots) staining present (Oxford scale)
  * Tear film break-up time (TBUT) less than or equal to 8 seconds
* Received study information and expressed willingness to take part in this study
* Confirmed able to attend the assessment visits described in the patient information
* Able and willing to complete the patient information diaries

Exclusion Criteria:

* Taking medication (except dry eye treatments) that is known to affect the tear film
* Currently using moisture chamber or goggles
* Active ocular surface pathology other than dry eye
* Ocular topography that in the clinician opinion would make OmniLenz BCL treatment inappropriate
* Allergic to ingredients within Omnigen (i.e. the antibiotics)
* History of:

  * Ocular herpetic keratitis
  * Ocular surgery in past 6 months
  * Use of glaucoma medicine
  * Surgery for glaucoma
* Eyelid abnormalities or extensive ocular scarring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Symptoms | 12 weeks post baseline
  Symptoms assessed with the Ocular Surface Disease Index questionnaire [0-100 range, higher worse]

SECONDARY OUTCOMES:
Change in Symptoms over time | 2, 4,12 and 24 weeks post baseline
  Change in the average Ocular Surface Disease Index score [0-100 range, higher worse]and its subscales at each time point versus baseline and control lens
Change in visual acuity over time | 2, 4, and 12 weeks post baseline
  Change in visual acuity (distance, best corrected) in logMAR notation with time versus baseline and control lens
Change in tear meniscus height over time | 2, 4, and 12 weeks post baseline
  Change in tear meniscus height (in mm) with time versus baseline and control lens
Change in non-invasive tear breakup time over time | 2, 4, and 12 weeks post baseline
  Change in non-invasive tear break-up time (in seconds, average of 3 reading) with time versus baseline and control lens
Change in ocular surface staining over time | 2, 4, and 12 weeks post baseline
  Change in corneal and conjunctival staining (number of punctate spots observed) with time versus baseline and control lens
Change in ocular redness over time | 2, 4, and 12 weeks post baseline
  Change in bulbar and limbal hyperaemia [Efron grade 0-4, lower number indicates less red] with time versus baseline and control lens
Health Utility | 24 weeks compared to baseline
  EQ-5D questionnaire [not an abbreviation; the 5 health states are report as the percent of participants reporting each level from 1-3 where lower is better health]

OTHER OUTCOMES:
Exploratory sampling/imaging - tear film | 2, 4 and 12 weeks post baseline
  Change in sampled tears (inflammatory marker presence) with time compared to baseline and control lens
Exploratory sampling/imaging - keratocytes | 2, 4 and 12 weeks post baseline
  Change in keratocyte like cells (number observed) on confocal imaging with time compared to baseline and control lens
Exploratory sampling/imaging - corneal nerves | 2, 4 and 12 weeks post baseline
  Change in corneal nerve density (area) on confocal imaging with time compared to baseline and control lens
Proportion of patients who find the treatment acceptable | 2 weeks of treatment
  Patients who are able to tolerate/complete at least 7 days of treatment
Use of concomitant medication | 4 and 12 weeks post-treatment compared to baseline
  Number of times artificial tear eye drops reported used

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hopkinson, PhD, Study Director — NuVision
Locations (1):
- Aston University, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized clinical data will be shared with other researchers on request.
Supporting Information: Study Protocol
Time Frame: After results publication
Access Criteria: Contact j.s.w.wolffsohn@aston.ac.uk

REFERENCES:
- [Background] McDonald MB, Sheha H, Tighe S, Janik SB, Bowden FW, Chokshi AR, Singer MA, Nanda S, Qazi MA, Dierker D, Shupe AT, McMurren BJ. Treatment outcomes in the DRy Eye Amniotic Membrane (DREAM) study. Clin Ophthalmol. 2018 Apr 9;12:677-681. doi: 10.2147/OPTH.S162203. eCollection 2018. PMID 29670328